CLINICAL TRIAL: NCT05033665
Title: The Impact of Adequate Water Intake on Exercise Performance and Mood in Women and Men
Acronym: WEXMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013646
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Dehydration; Mood
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euhydrated (Active Comparator): Afternoon urine osmolality < 800 mmol/kg or urine specific gravity < 1.020.
  Interventions: Behavioral: Maintain adequate water consumption
- Underhydrated (Experimental): Afternoon urine osmolality ≥ 800 mmol/kg or urine specific gravity ≥ 1.020.
  Interventions: Behavioral: Increase water consumption

INTERVENTIONS:
Behavioral: Increase water consumption — The underhydrated individuals will be instructed to increase their water intake for one week in order to meet the following two criteria: a) urinate at least 7 times per day and b) have straw-like color urine. A 2-mile run will be completed before and after the 7-day intervention.
  Arms: Underhydrated
Behavioral: Maintain adequate water consumption — The subjects that are classified as euhydrated will be asked to maintain high water intake for one week to ensure proper hydration. A 2-mile run will be completed before and after the 7-day intervention.
  Arms: Euhydrated

SUMMARY:
Dehydration is defined as the state of water deficit due to excessive water losses and/or small water intake. Underhydration is the result of inadequate water intake leading to activation of water hormonal homeostasis, characterized by elevated vasopressin, lower urinary output, and concentrated urine without any measurable changes in total body water. It is well established that dehydration (water deficit) decreases exercise performance and worsens mood, mainly in women. However, the impact of increased water intake in underhydrated individuals on their exercise capacity and mood is not known.

The aim of the proposed study is to investigate the impact of increased water intake in underhydrated individuals on aerobic exercise performance and mood in both women and men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Residence in Arizona

Exclusion Criteria:

* Use of diuretics
* Use of anti-depressive medication
* Current pregnancy or lactation
* Current use of injectable insulin
* Diagnosed with irritable bowel syndrome
* Do not pass the Physical Activity Readiness Questionnaire for Everyone (PAR-Q) screening

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
2-mile run-time (min) | Day 1
2-mile run-time (min) | Day 8
Mood | Pre-trial on day 1
  Profile of Mood States questionnaire (POMS 2®-Adult Short, Multi-Health Systems Inc.)
Mood | Post-trial on day 1
  Profile of Mood States questionnaire (POMS 2®-Adult Short, Multi-Health Systems Inc.)
Mood | Pre-trial on day 8
  Profile of Mood States questionnaire (POMS 2®-Adult Short, Multi-Health Systems Inc.)
Mood | Post-trial on day 8
  Profile of Mood States questionnaire (POMS 2®-Adult Short, Multi-Health Systems Inc.)
Urine osmolality (mmol/kg) | 4 - 8 PM on day 0
Urine osmolality (mmol/kg) | 4 - 8 PM on day 7
Urine osmolality (mmol/kg) | Upon waking (first morning sample) on day 1
Urine osmolality (mmol/kg) | Upon waking (first morning sample) on day 8
Urine specific gravity | 4 - 8 PM on day 0
Urine specific gravity | 4 - 8 PM on day 7
Urine specific gravity | Upon waking (first morning sample) on day 1
Urine specific gravity | Upon waking (first morning sample) on day 8

SECONDARY OUTCOMES:
Urine color | 4 - 8 PM on day 0
  Armstrong validated 8-color scale. Minimum score: 1. Maximum score: 8. A higher score indicates a worse outcome (e.g., dehydrated).
Urine color | 4 - 8 PM on day 7
  Armstrong validated 8-color scale. Minimum score: 1. Maximum score: 8. A higher score indicates a worse outcome (e.g., dehydrated).
Urine color | Upon waking (first morning sample) on day 1
  Armstrong validated 8-color scale. Minimum score: 1. Maximum score: 8. A higher score indicates a worse outcome (e.g., dehydrated).
Urine color | Upon waking (first morning sample) on day 8
  Armstrong validated 8-color scale. Minimum score: 1. Maximum score: 8. A higher score indicates a worse outcome (e.g., dehydrated).
Thirst perception | 4 - 8 PM on day 0
  175 mm visual analog scale. Minimum score: 0 (not thirsty at all). Maximum score: 175 (extremely thirsty). A higher score indicates a worse outcome (e.g., more thirsty).
Thirst perception | 4 - 8 PM on day 7
  175 mm visual analog scale. Minimum score: 0 (not thirsty at all). Maximum score: 175 (extremely thirsty). A higher score indicates a worse outcome (e.g., more thirsty).
Thirst perception | Upon waking (first morning sample) on day 1
  175 mm visual analog scale. Minimum score: 0 (not thirsty at all). Maximum score: 175 (extremely thirsty). A higher score indicates a worse outcome (e.g., more thirsty).
Thirst perception | Upon waking (first morning sample) on day 8
  175 mm visual analog scale. Minimum score: 0 (not thirsty at all). Maximum score: 175 (extremely thirsty). A higher score indicates a worse outcome (e.g., more thirsty).

CONTACTS AND LOCATIONS:
Locations (1):
- Interdisciplinary Science and Technology Building 8, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No